CLINICAL TRIAL: NCT05619406
Title: Systematic Investigation of Blacks With Stroke - GENOMICS (SIBS-GENOMICS)
Brief Title: Systematic Investigation of Blacks With Stroke - GENOMICS
Acronym: SIBSGENOMICS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Hospital, Ibadan (Other)
Collaborators: Medical University of South Carolina (Other); University of Ibadan (Other); Federal Medical Centre, Abeokuta (Unknown); Ahmadu Bello University Teaching Hospital (Other); Bayero University Kano, Nigeria (Other); Kwame Nkrumah University of Science and Technology (Other); Korle-Bu Teaching Hospital, Accra, Ghana (Other); University of Alabama at Birmingham (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Mayowa Owolabi, Professor, University College Hospital, Ibadan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UI/EC/18/0706
Record Dates: First submitted 2022-10-24; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Hypertension; Adult; Dyslipidemias; Physical Inactivity; Diabetes; Alcohol Consumption
Keywords: Stroke-free adults; Riskometer App; Africans
MeSH Terms: conditions — Hypertension; Dyslipidemias; Sedentary Behavior; Diabetes Mellitus; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: The relational data model is adopted in the Model component of the system
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and outcome assessor will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): The Control Group will be screened at baseline and be informed of their risk factors. They will be counselled to consult their provider following baseline risk factor assessment but this advice will not be reinforced by exposure to the app, stroke video, or module content. At the end of the study (EOS), they will complete a questionnaire to assess possible contamination with the intervention.
  Interventions: Device: Riskometer Application
- Intervention (Experimental): The riskometer app will be administered one-on-one to the participants using a smartphone and eventually score and assess them using the global risk score
  Interventions: Behavioral: Routine Clinic Therapy

INTERVENTIONS:
Device: Riskometer Application — The intervention group participants at baseline will be assessed by installing a riskometer app on their mobile phones to calculate their global stroke risk score. They will be shown their risk scores and the specific risk factors identified through the screening. They will be counselled and supported to manage their risk factors through lifestyle changes and visit their healthcare provider for appropriate care.
  Arms: Control
Behavioral: Routine Clinic Therapy — After their assessment by the blinded adjudicator, the controls will visit the study doctor to obtain the routine clinic therapy and then will be allowed to go home.
  Arms: Intervention

SUMMARY:
The overall goal of SIBS-GENOMICS is to utilize the best available contextual data on stroke in Africa to develop & validate stroke risk estimation models, translate the best model into a mobile phone app and conduct a randomized control trial of the app with a co-created motivational education video, to determine their effectiveness for improvement of stroke risk factor awareness and global risk reduction among Africans.

DETAILED DESCRIPTION:
Africa now bears a foremost burden of stroke worldwide with age standardized stroke incidence rate of up to 316 per 100,000, a prevalence of 1.46 per 1,000 population,1 month fatality of 40% & a 3-year mortality rate of 84%.

The burden of stroke on the continent falls heavily on the young productive age group & is associated with profound diminution in the quality of life via disability, depression, & vascular cognitive impairment.

World Health Organization estimates that stroke deaths in LMIC account for 86% of stroke deaths worldwide & disability-adjusted life years lost in LMIC is 7X those lost in high-income countries (HIC). Beyond the personal toll, costs related to stroke are prohibitive and threaten to erode the recent economic gains in Africa where the stroke is a major threat to brain health, brain capital and human capital. The surge in stroke burden in Africa is driven by an unprecedented rise in precursory modifiable cardiometabolic risk factors.

There is an urgent need to deploy evidence-based approaches using the best available context-specific data to surmount the stroke epidemic on the continent by developing population-wide preventive interventions. Achieving this goal requires tackling key barriers to stroke prevention such as lack of awareness and self-directed action to control its risk factors.

Systematic Investigation of Blacks With Stroke (SIBS-GENOMICS) is poised to utilize the best available context-specific data on stroke in Africa to improve, validate, and co-create the first ever Afrocentric stroke riskometer mobile phone application, a self-management tool for stroke prevention. The app, along with a tailored co-created stroke prevention motivational video and educational modules with customized behavioral change activities, will be evaluated for effectiveness to improve individual stroke risk factor awareness and control in the first-of-its-kind randomized control trial (RCT) for a digital tool for primary stroke prevention in Africa.

With the scarcity of acute care and rehabilitation services, coupled with the chronic economic burden imposed by stroke, prevention is evidently the best option towards reducing its burden in Africa. This is concordant with the core mission of the NINDS to reduce the burden of stroke in the USA and globally through translational research and innovation.

ELIGIBILITY:
Inclusion Criteria:

* male or female (sex is a biologic variable of interest).
* age greater than or equal to 18 years.
* with at least 2 stroke risk factors based on the list of 11 top most modifiable risk factors identified in the SIREN study (including hypertension, diabetes mellitus, dyslipidemia, smoking, overweight, physical inactivity, or unbalanced/poor diet).
* ownership or access to smartphones in consenting stroke-free adults.

Exclusion Criteria:

* prior history of vascular disease (e.g., stroke, transient ischemic attack, angina, myocardial infarction, peripheral vascular disease, and atrial fibrillation), or cognitive impairment; not comfortable reading and writing, depression or other psychiatric disorders (through personal declaration) likely to affect the interventions; participation in another RCT; other conditions rendering the individual unsuitable to participate in this research as judged by treating physicians.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-20 (Actual); Primary Completion 2022-11-06 (Actual); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 2 months
  Total stroke risk probability (0 to 100%) calculated by the software. Reduction in total score of at least 10% over 2 months

SECONDARY OUTCOMES:
Secondary Outcome | 2 months
  Stroke risk factors awareness score. List of risk factors will be based on SIREN findings and developed into a questionnaire which will be pretested and validated; and translated/back-translated. Change in individual risk factors will also be assessed and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Mayowa O. Owolabi, MD, Principal Investigator — College of Medicine University of Ibadan; Bruce Ovbiagele, MD, Principal Investigator — University of California, San Francisco; Fred S. Sarfo, PhD, Principal Investigator — Kwame Nkrumah University of Science & Technology (KNUST); Benjamin S. Aribisala, PhD, Principal Investigator — Lagos State University, (LASU); Michelle Nichols, PhD, Principal Investigator — Medical University of South Carolina; Oyedunni S. Arulogun, PhD, Principal Investigator — University of Ibadan; Carolyn Jenkins, PhD, Principal Investigator — Medical University of South Carolina; Bukola Ajala, PhD, Principal Investigator — University of Ibadan; Onoja M. Akpa, PhD, Principal Investigator — University of Ibadan; Odun J. Akinyemi, PhD, Principal Investigator — University of Ibadan; Rufus A. Akinyemi, PhD, Principal Investigator — University of Ibadan; Reginald O. Obiako, PhD, Principal Investigator — Ahmadu Bello University Teaching Hospital, (ABUTH) Zaria
Locations (3):
- Kwame Nkrumah University of Science and Technology (KNUST), Kumasi, Ghana
- Nigeria (2):
  - Ahmadu Bello University Teaching Hospital, (ABUTH) Zaria, Zaria, Kaduna State
  - University College Hospital, Ibadan, Oyo State

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarfo FS, Akinyemi JO, Obiako R, Nichols M, Fakunle AG, Adusei N, Ampofo M, Arulogun O, Jenkins C, Akpa OM, Aribisala B, Abdulrasaq S, Akinyemi R, Ovbiagele B, Owolabi MO. Effect of an Educational Intervention for Primary Stroke Risk Reduction in Ghana and Nigeria: Pilot Randomized Controlled Trial. Stroke. 2023 Jun;54(6):1660-1664. doi: 10.1161/STROKEAHA.123.042618. Epub 2023 May 4. PMID 37139815

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-09-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT05619406/Prot_ICF_000.pdf